CLINICAL TRIAL: NCT00604279
Title: A Randomized, Open-Label, Parallel Group Comparative Study of Paliperidone Palmitate (50, 100, 150 mg eq) and Risperidone LAI (25, 37.5, or 50 mg) in Subjects With Schizophrenia
Brief Title: A Comparative Study of Paliperidone Palmitate and Risperidone Long Acting Injection (LAI) in Participants With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013150; R092670PSY3008
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone; Paliperidone palmitate; Risperidone; Risperidone long acting injection; R092670
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paliperidone palmitate (Experimental): Paliperidone palmitate suspension for intramuscular injection at a dose of 150 milligram equivalent (mg eq.) at baseline, 100 mg eq. on Day 8, flexible dose, either 50 or 100 mg eq on Day 36 and 50, 100, or 150 mg eq.on Day 64 depending on investigator's discretion.
  Interventions: Drug: Paliperidone palmitate (R092670)
- Risperidone long acting injection (LAI) (Active Comparator): Risperidone LAI intramuscular at a dose of 25 milligram (mg) on Day 8 and Day 22; flexible dose of either 25 or 37.5 mg on Day 36 with same dose on Day 50; and either 25, 37.5, or 50 mg on Day 64 with same dose on Day 78; along with oral risperidone 2 mg tablet on Day 1, flexible doses (1-6 mg/day) for first 28 days; and 1-2 mg/day during Day 36-57 and Day 64-85 if the dose of risperidone LAI was increased on Day 36 and Day 64.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Paliperidone palmitate (R092670) — Paliperidone palmitate suspension for intramuscular injection at a dose of 150 milligram equivalent (mg eq.) at baseline, 100 mg eq. on Day 8, flexible dose, either 50 or 100 mg eq on Day 36 and 50, 100, or 150 mg eq.on Day 64 depending on investigator's discretion.
  Arms: Paliperidone palmitate
Drug: Risperidone — Risperidone LAI intramuscular at a dose of 25 mg on Day 8 and Day 22; flexible dose of either 25 or 37.5 mg on Day 36 with same dose on Day 50; and either 25, 37.5, or 50 mg on Day 64 with same dose on Day 78; along with oral risperidone 2 mg tablet on Day 1, flexible doses (1-6 mg/day) for first 28 days; and 1-2 mg/day during Day 36-57 and Day 64-85 if the dose of risperidone LAI was increased on Day 36 and Day 64.
  Arms: Risperidone long acting injection (LAI)

SUMMARY:
The purpose of this study is to compare the efficacy of paliperidone palmitate and risperidone long acting injection (LAI) in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) along with safety and tolerability.

DETAILED DESCRIPTION:
This is a randomized (assigned by chance), open-label (all people know the identity of the intervention), active-controlled, parallel-group (a medical research study comparing the response in two or more groups of participants receiving different treatments), multicenter (when more than one hospital or medical school team work on a medical research study) comparative study in participants with schizophrenia. This study comprises a screening period of not more than 7 days and a 13-week open-label treatment period. Paliperidone palmitate will be administered as intramuscular injection (injection of a substance into a muscle) of 150 milligram equivalent (mg eq.) at baseline, 100 mg eq. at Day 8, flexible dose on Day 36 (50 or 100 mg eq.) and on Day 64 (50, 100 or 150 mg eq.) depending on investigator's discretion. Risperidone LAI will be administered at a dose of 25 mg at Day 8 and Day 22, flexible dose on Day 36 (25 or 37.5 mg) and Day 64 (25, 37.5, or 50 mg). Dose on Day 50 is the same as Day 36 and dose on Day 78 is the same as Day 64. Participants will receive oral risperidone tablets (1 to 6 mg/day) for the first 4 weeks of the open-label treatment period. Each participant may receive oral risperidone tablets (1 to 2 mg daily) for up to 3 weeks at Day 36 and Day 64 if the dose of risperidone LAI was increased on Day 36 and Day 64. Efficacy will primarily be assessed using the Positive and Negative Syndrome Scale (PANSS). Participants' safety will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet diagnostic criteria for schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) (disorganized type [295.10], catatonic type [295.20], paranoid type [295.30], residual type [295.60], or undifferentiated type [295.90]) for at least 1 year before screening and prior medical records, written documentation, or verbal information obtained from previous psychiatric providers obtained by the investigator must be consistent with the diagnosis of schizophrenia
* A total Positive and Negative Syndrome Scale (PANSS) score between 60 and 120, inclusive, at screening and baseline
* Body mass index (BMI) of equal to or greater than 17.0 kilogram per meter square (kg/m^2)
* Female participants must be postmenopausal for at least 2 years, surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control before study entry and throughout the study
* Be capable of self-administering study medication (applies to oral supplementation) or have assistance with study medication administration consistently available throughout the first 4 weeks of the study Exclusion Criteria:
* A primary, active DSM-IV diagnosis on Axis I other than schizophrenia
* A decrease of at least 25 percent in the total PANSS score between screening and baseline
* Participants who have previously participated in this study
* A DSM-IV diagnosis of active substance dependence within 3 months before screening (nicotine and caffeine are not exclusionary)
* History of treatment resistance as defined by failure to respond to 2 adequate treatments with different antipsychotic medications (an adequate treatment is defined as a minimum of 6 weeks at maximum tolerated dosage)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd. Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (8):
- China (8):
  - Baoding
  - Beijing
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai
  - Wuhan
  - Xi'an

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone Palmitate: Paliperidone palmitate (R092670) suspension for intramuscular (directly into a muscle) injection at a dose of 150 milligram equivalent (mg eq.) at baseline, 100 mg eq. on Day 8, flexible dose, either 50 or 100 mg eq on Day 36 and 50, 100, or 150 mg eq. on Day 64 depending on investigator's discretion.
Period: Overall Study
Arm/Group | Paliperidone Palmitate | Risperidone Long Acting Injection (LAI)
Started | 229 | 223
Completed | 165 | 185
Not Completed | 64 | 38
Not completed — Lack of Efficacy | 22 | 9
Not completed — Lost to Follow-up | 9 | 14
Not completed — Pregnancy | 2 | 0
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 16 | 5
Not completed — Adverse Event | 4 | 5
Not completed — Other | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Paliperidone Palmitate: Paliperidone palmitate suspension for intramuscular injection at a dose of 150 milligram equivalent (mg eq.) at baseline, 100 mg eq. on Day 8, flexible dose, either 50 or 100 mg eq on Day 36 and 50, 100, or 150 mg eq. on Day 64 depending on investigator's discretion.
- Total: Total of all reporting groups
Arm/Group | Paliperidone Palmitate | Risperidone Long Acting Injection (LAI) | Total
Number analyzed (Participants) | 229 | 223 | 452
Age Continuous [Mean (Standard Deviation); unit: years] | 32 (10.75) | 31.5 (11.03) | 31.7 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 129 | 271
  Male | 87 | 94 | 181
Age Categorical [Number; unit: Participants]
  18-25 Years | 87 | 92 | 179
  26-50 Years | 125 | 114 | 239
  51-65 Years | 17 | 17 | 34
  >65 Years | 0 | 0 | 0
  <18 Years | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Day 92 or Early Withdrawal
Description: The PANSS provides a total score (sum of the scores of all 30 items) and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 (absent) to 210 (extreme psychopathology). Higher change scores indicate worsening.
Time Frame: Baseline, Day 92 or early withdrawal
Population: Per Protocol Analysis Set included participants who received at least 2 injections of study medication had minimum 5 weeks of exposure to study treatment; had baseline and at least 1 post randomization measurement for primary efficacy variable and who did not have major protocol violations.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Paliperidone Palmitate | Risperidone Long Acting Injection (LAI)
Number analyzed (Participants) | 205 | 208
Units on scale
  Baseline | 82.1 (11.95) | 84.4 (12.69)
  Change at Day 92 or Early Withdrawal | -23.6 (16.28) | -26.9 (15.43)
Statistical Analysis 1: Comparison: Paliperidone Palmitate vs Risperidone Long Acting Injection (LAI); Test type: Non-Inferiority or Equivalence — The predetermined margin for non-inferiority of paliperidone palmitate was 5.5 points; ANCOVA; Analysis of covariance (ANCOVA) model with treatment as a factor, and baseline value as a covariate was used; Least Square Mean Difference = -2.3, 95% CI [-5.20 to 0.63], Standard Error of Mean 1.48

2. Secondary Outcome: Change From Baseline in Personal and Social Performance (PSP) Score at Day 92 or Early Withdrawal
Description: This PSP assesses the degree of a participant's dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate the degree of difficulty (1, absent to 4, very severe) in each of the 4 domains. Based on the four domains there will be one total score. Participants with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; <= 30, functioning so poorly as to require intensive supervision.
Time Frame: Baseline, Day 92 or early withdrawal
Population: Per Protocol Analysis Set. Here "N" (Number of Participants Analyzed) represents number of participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Paliperidone Palmitate | Risperidone Long Acting Injection (LAI)
Number analyzed (Participants) | 184 | 190
Units on scale
  Baseline | 47.8 (12.42) | 45.3 (11.29)
  Change at Day 92 or Early Withdrawal | 16.8 (14.76) | 18.6 (13.92)
Statistical Analysis 1: Comparison: Paliperidone Palmitate vs Risperidone Long Acting Injection (LAI); Test type: Superiority or Other; ANCOVA; Analysis of covariance (ANCOVA) model with treatment as a factor, and baseline value as a covariate was used; Least Square Mean Difference = 0.5, 95% CI [-2.14 to 3.12], Standard Error of Mean 1.34

3. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score at Day 92 or Early Withdrawal
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher change scores indicate worsening.
Time Frame: Baseline, Day 92 or early withdrawal
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Paliperidone Palmitate | Risperidone Long Acting Injection (LAI)
Number analyzed (Participants) | 204 | 207
Units on scale
  Baseline | 4.9 (0.82) | 5.0 (0.81)
  Change at Day 92 or Early Withdrawal | -1.5 (1.24) | -1.7 (1.16)
Statistical Analysis 1: Comparison: Paliperidone Palmitate vs Risperidone Long Acting Injection (LAI); Test type: Superiority or Other; ANCOVA; Analysis of covariance (ANCOVA) model with treatment as a factor, and baseline value as a covariate was used; Least Square Mean Difference = -0.1, 95% CI [-0.33 to 0.10], Standard Error of Mean 0.11

4. Secondary Outcome: Change From Baseline in the Sleep Visual Analog Scale (VAS) Score at Day 92 or Early Withdrawal
Description: The self-administered sleep VAS scale (0-100 millimeter [mm]) rates quality of sleep (QoS) and daytime drowsiness (DD). Participants indicate mark on the scale to represent how well they have slept in the previous 7 days, score ranges from 0 mm (very badly) to 100 mm (very well); and how often they have felt drowsy within the previous 7 days, from 0 mm (not at all) to 100 mm (all the time).
Time Frame: Baseline, Day 92 or early withdrawal
Population: Per Protocol Analysis Set.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Paliperidone Palmitate | Risperidone Long Acting Injection (LAI)
Number analyzed (Participants) | 205 | 208
millimeter (mm)
  QoS, Baseline | 64.1 (25.40) | 66.6 (24.22)
  QoS, Change at Day 92 or Early Withdrawal | 8.2 (26.95) | 10.0 (26.18)
  DD, Baseline | 29.9 (25.25) | 29.6 (23.50)
  DD, Change at Day 92 or Early Withdrawal | -4.1 (27.26) | -4.9 (24.12)
Statistical Analysis 1: Comparison: Paliperidone Palmitate vs Risperidone Long Acting Injection (LAI); Statistical Analysis for Quality of sleep; Test type: Superiority or Other; ANCOVA; Analysis of covariance (ANCOVA) model with treatment as a factor, and baseline value as a covariate was used; Least Square Mean Difference = 3.4, 95% CI [-0.67 to 7.50], Standard Error of Mean 2.08
Statistical Analysis 2: Comparison: Paliperidone Palmitate vs Risperidone Long Acting Injection (LAI); Statistical Analysis for Daytime drowsiness; Test type: Superiority or Other; ANCOVA; Analysis of covariance (ANCOVA) model with treatment as a factor, and baseline value as a covariate was used; Least Square Mean Difference = -1.1, 95% CI [-5.04 to 2.90], Standard Error of Mean 2.02

5. Secondary Outcome: Percentage of Participants Who Responded to PANSS Total Score at Day 92 or Early Withdrawal
Description: A responder is defined as a participant who improved from baseline in the PANSS total score by 30 percent or more.
Time Frame: Day 92 or early withdrawal
Population: Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Paliperidone Palmitate | Risperidone Long Acting Injection (LAI)
Number analyzed (Participants) | 205 | 208
Percentage of participants | 70.7 (25.40) | 78.4 (24.22)
Statistical Analysis 1: Comparison: Paliperidone Palmitate vs Risperidone Long Acting Injection (LAI); Test type: Superiority or Other; Cochran-Mantel-Haenszel; Point estimate of relative risk = 0.9, 95% CI [0.81 to 1.01]

ADVERSE EVENTS:
Arm/Group | Paliperidone Palmitate | Risperidone Long Acting Injection (LAI)
Serious Adverse Events (participants affected / at risk) | 3/229 | 8/223
Other Adverse Events (participants affected / at risk) | 115/229 | 127/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Palmitate (N=229) | Risperidone Long Acting Injection (LAI) (N=223)
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Psychiatric symptom (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Refusal of treatment by patient (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Palmitate (N=229) | Risperidone Long Acting Injection (LAI) (N=223)
Constipation (Gastrointestinal disorders) | 17 | 12
Upper respiratory tract infection (Infections and infestations) | 18 | 13
Blood prolactin increased (Investigations) | 17 | 12
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 10 | 16
Akathisia (Nervous system disorders) | 30 | 44
Bradykinesia (Nervous system disorders) | 16 | 9
Tremor (Nervous system disorders) | 24 | 40
Anxiety (Psychiatric disorders) | 10 | 13
Insomnia (Psychiatric disorders) | 41 | 30
Restlessness (Psychiatric disorders) | 16 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to publication and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The paper that incorporates confidential information requires Sponsor's written consent. PI will withhold publication for up to an additional 60 days to allow for filing of a patent application.